CLINICAL TRIAL: NCT03981380
Title: 11C-PIB PET Study in the Multi Ethnic Study of Atherosclerosis at Columbia University
Brief Title: 11C-PIB PET Study in MESA at Columbia University
Status: Completed | Type: Observational
Sponsor: José A. Luchsinger (Other)
Collaborators: Wake Forest University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, José A. Luchsinger, Associate Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Other Study IDs: AAAS2808; R01AG058969 (NIH)
Record Dates: First submitted 2019-06-07; First posted 2019-06-10 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Cognitive Impairment; Vascular Diseases; Alzheimer Disease; Atherosclerosis
Keywords: Alzheimer Disease; Cognitive Impairment; 11C-PiB; Atherosclerosis
MeSH Terms: conditions — Cognitive Dysfunction; Vascular Diseases; Alzheimer Disease; Atherosclerosis | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will store plasma and serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MESA study participants: Current participants in the MESA study in New York City, 60 years or older, fluent in English or Spanish, able to participate in the brain imaging study
  Interventions: Drug: 11C-PIB

INTERVENTIONS:
Drug: 11C-PIB — Participants will be injected with an intravenous bolus of up to 5-15mCi (370 MBq) (+/-10%) of [11C]PiB (over 5-10 seconds).
  Other Names: PIB

SUMMARY:
The investigators will conduct a study of brain positron emission tomography (PET) using 11C-PIB for the imaging of brain amyloid in 250 participants in the Multiethnic study of atherosclerosis (MESA) at Columbia University Irving Medical Center in New York City. Participants will be imaged only once with Pittsburgh Compound B (PIB) PET.

DETAILED DESCRIPTION:
This is a single center PET study of 11C-PIB. Eligible participants are current participants in the MESA study in New York City, without contraindications to MRI or PET procedures. Those eligible will have one brain PET scan with 11C-PIB within 12 months of a brain MRI. Vital signs will be checked prior to injection of 11C-PIB, 10 minutes after the injection, and again at the completion of the PET scan. The primary outcome measure for amyloid will be whole brain 11C-PIB SUVR. The relation between exposure groups and amyloid in the brain will be analyzed using linear regression.

ELIGIBILITY:
Inclusion Criteria:

* Current participants in MESA study at Columbia University
* 60 years or older
* Fluent in English and/or Spanish.
* Able to participate in all scheduled evaluations and to complete all required tests and procedures.

Exclusion Criteria:

* Active treatment for cancer
* Any serious medical condition which would prevent long-term participation
* Pregnancy
* Weight >300 pounds
* Participants previously diagnosed or adjudicated to have dementia
* Participants unwilling to undergo cognitive testing
* Plans to leave the community within five years
* Language barrier (speaks other than English, Spanish, Chinese)
* Inability to give informed consent or to obtain consent from a Legally Authorized Representative (LAR)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Current participants in MESA study in New York City
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Whole Brain 11C-PIB SUVR | 40 to 90 minutes post injection
  Standardized uptake value ratio (SUVR) of 11C-PIB;The extent of Aβ deposition in the brain will be quantified by[11C]PiB uptake visualized by PET using standardized uptake volume ratio (SUVR) of 6 primary cortical areas (i.e., anterior cingulate, prefrontal cortex, lateral temporal cortex, posterior parietal cortex, precuneus cortex, and anteroventral striatum) relative to the uptake in the cerebellum

CONTACTS AND LOCATIONS:
Overall Officials: José Luchsinger, MD, MPH, Principal Investigator — Professor of Medicine and Epidemiology
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) may be shared at the end of data collection with a mechanism supported by the National Institute on Aging